CLINICAL TRIAL: NCT02333331
Title: A 28 Week, Randomized, Double-blind, Placebo-controlled, Two-part, Multi-center, Parallel Group Dose Range Finding Study to Assess the Effect of Monthly Doses of Bimagrumab 70, 210, and 700 mg on Skeletal Muscle Strength and Function in Older Adults With Sarcopenia (InvestiGAIT)
Brief Title: Dose Range Finding Study of Bimagrumab in Sarcopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBYM338E2202
Record Dates: First submitted 2014-12-10; First posted 2015-01-07 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-07

CONDITIONS: Sarcopenia
Keywords: Sarcopenia, muscle wasting, elderly, strength, physical function, muscle, gait speed
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy | interventions — bimagrumab; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BYM338 70 mg (Experimental): BYM338 70 mg intravenous infusion
  Interventions: Drug: bimagrumab
- BYM338 210 mg (Experimental): BYM338 210 mg intravenous infusion
  Interventions: Drug: bimagrumab
- BYM338 700 mg (Experimental): BYM338 700 mg intravenous infusion
  Interventions: Drug: bimagrumab
- Placebo (Placebo Comparator): Placebo intravenous infusion
  Interventions: Other: placebo

INTERVENTIONS:
Drug: bimagrumab — Bimagrumab will be administered as an intravenous infusion starting on Day 1 until week 21.
  Other Names: BYM338
  Arms: BYM338 210 mg; BYM338 70 mg; BYM338 700 mg
Other: placebo — Placebo will be administered as an intravenous infusion starting on Day 1 until week 21.
  Other Names: 5% dextrose
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the efficacy of repeat dosing with multiple dose levels of bimagrumab on patient physical function, skeletal muscle mass and strength in older adults with sarcopenia. In addition, this study generated data on the safety, tolerability, and pharmacokinetics of bimagrumab in older adults with sarcopenia.

ELIGIBILITY:
Inclusion Criteria:

* Low muscle mass as confirmed by DXA;
* Low gait speed <0.8 m/s
* SPPB score less than or equal to 9;
* Weigh at least 35 kg;
* Adequate dietary intake;

Exclusion Criteria:

* A lower limb fracture in the past 6 months or any impairment or disease severely affecting gait (e.g. stroke with hemiparesis, myasthenia gravis, Parkinson's disease, peripheral polyneuropathy, intermittent claudication in advanced peripheral vascular disease, spinal stenosis, or severe osteoarthritis of the knee or hip with ineffective pain management);
* Requires regular assistance from another person for general activities of daily living (e.g. bathing, dressing, toileting).
* Intraocular surgery and laser procedures for refractive correction within 6 months prior to screening;
* Any underlying muscle disease including active myopathy or muscular dytrophy;
* Confirmed diagnosis of heart failure classified as New York Heart Association Class III or IV (e.g. dilated cardiomyopathy);
* Type I diabetes or uncontrolled Type 2 diabetes;
* Chronic kidney disease [estimated glomerular filtration rate (GFR) < 30 mL/min];
* History of confirmed chronic obstructive pulmonary disease with a severity grade > 2 on the Medical Research Council Dyspnea Scale;
* Confirmed rheumatoid arthritis or other systemic autoimmune disease requiring immunosuppressive therapy or corticosteroids >10 mg/d prednisone equivalent;
* Known history or presence of severe active acute or chronic liver disease (e.g., cirrhosis);
* Myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention (e.g. angioplasty or stent placement), or deep vein thrombosis/pulmonary embolism within 12 weeks of screening;
* Active cancer (i.e., under current treatment), or cancer requiring treatment in the last 5 years excluding non-melanoma skin cancers or cancers with excellent prognosis (e.g., early stage prostate or breast cancer, carcinoma in situ of the uterine cervix);
* Any chronic active infection (e.g., HIV, Hepatitis B or C, tuberculosis, etc).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (17):
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Cypress, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Farmington, Connecticut
  - Novartis Investigative Site, Gainesville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Miami Lakes, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Gainesville, Georgia
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Madison, Wisconsin
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, St Albans, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Opava
  - Novartis Investigative Site, Prague
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Copenhagen NV
- France (4):
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Würzburg
- Japan (12):
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Mizunami, Gifu
  - Novartis Investigative Site, Nara, Nara
  - Novartis Investigative Site, Kawachi-Nagano, Osaka
  - Novartis Investigative Site, Kitaadachigun Inamachi, Saitama
  - Novartis Investigative Site, Kitamoto, Saitama
  - Novartis Investigative Site, Yoshinogawa, Tokushima
  - Novartis Investigative Site, Itabashi Ku, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Koto-ku, Tokyo
  - Novartis Investigative Site, Musashimurayama, Tokyo
- Russia (3):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
- South Korea (3):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
- Spain (4):
  - Novartis Investigative Site, Albacete, Castille-La Mancha
  - Novartis Investigative Site, Getafe, Madrid
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Basel, CH
  - Novartis Investigative Site, Geneva
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Rooks D, Swan T, Goswami B, Filosa LA, Bunte O, Panchaud N, Coleman LA, Miller RR, Garcia Garayoa E, Praestgaard J, Perry RG, Recknor C, Fogarty CM, Arai H, Chen LK, Hashimoto J, Chung YS, Vissing J, Laurent D, Petricoul O, Hemsley S, Lach-Trifilieff E, Papanicolaou DA, Roubenoff R. Bimagrumab vs Optimized Standard of Care for Treatment of Sarcopenia in Community-Dwelling Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2020836. doi: 10.1001/jamanetworkopen.2020.20836. PMID 33074327
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 220 patients were randomized to receive six doses of either BYM338 70 mg, BYM338 210 mg, BYM338 700 mg or the placebo. However, only 217 patients were enrolled and dosed with BYM338 or placebo due to the withdrawal of three patients who did not meet the inclusion/exclusion criteria prior to receiving the first dose.
Period: Overall Study
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo
Started | 19 | 18 | 113 | 67
Completed | 17 | 12 | 95 | 64
Not Completed | 2 | 6 | 18 | 3
Not completed — Adverse Event | 1 | 0 | 4 | 1
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 3 | 2 | 1
Not completed — Patient/Guardian Decision | 1 | 2 | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo | Total
Number analyzed (Participants) | 19 | 18 | 113 | 67 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.3 (5.89) | 78.0 (6.38) | 79.5 (5.46) | 78.3 (5.03) | 79.0 (5.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 66 | 43 | 126
  Male | 10 | 10 | 47 | 24 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 5 | 3 | 17 | 11 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 3 | 0 | 0 | 1 | 4
  White | 11 | 14 | 93 | 54 | 172
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Short Physical Performance Battery (SPPB) Score to Week 25
Description: Change from Baseline in total Short Physical Performance Battery (SPPB) Score to week 25; SPPB is a series of six activities involving three domains of physical function - balance, usual walking speed and rising from a chair , is commonly used globally to assess and quantify (score 0-12) lower extremity function and has been shown to predict future adverse health events. A decline of one or more points in the SPPB total score is predictive of a decrease in lower extremity function and future adverse clinical outcomes in older adults, including falls, hospitalizations, institutionalization, incident disability and death
Time Frame: Baseline, week 25
Population: Full Analysis Set (FAS) -comprised all patients to whom study treatment had been assigned. Following the intent to treat principle, patients were analyzed according to treatment assigned at randomization.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo
Number analyzed (Participants) | 19 | 18 | 113 | 67
Score on a scale
  Baseline: number analyzed (Participants) | 17 | 10 | 94 | 62
  Baseline | 7.1 (2.12) | 7.3 (2.11) | 7.2 (1.63) | 7.3 (1.67)
  Week 25: number analyzed (Participants) | 17 | 10 | 94 | 62
  Week 25 | 8.5 (2.48) | 8.7 (1.64) | 8.7 (2.12) | 8.4 (2.25)
Statistical Analysis 1: Comparison: BYM338 70 mg vs Placebo; Test type: Superiority; p = 0.274, Mixed Models Analysis; Mean Difference (Final Values) = 0.28, 95% CI 2-sided [-0.64 to 1.21]
Statistical Analysis 2: Comparison: BYM338 210 mg vs Placebo; Test type: Superiority; p = 0.320, Mixed Models Analysis; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [-0.83 to 1.35]
Statistical Analysis 3: Comparison: BYM338 700 mg vs Placebo; Test type: Superiority; p = 0.134, Mixed Models Analysis; Mean Difference (Final Values) = 0.31, 95% CI 2-sided [-0.24 to 0.87]

2. Secondary Outcome: Change From Baseline at Week 25 in the 6 Minute Walk Test (6MWT) Distance
Description: Change from Baseline at Week 25 in the 6 minute walk test (6MWT) distance to measure improvement in physical function
Time Frame: Baseline, week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo
Number analyzed (Participants) | 19 | 18 | 113 | 67
meters
  Baseline: number analyzed (Participants) | 19 | 18 | 112 | 67
  Baseline | 293.30 (91.842) | 291.81 (82.527) | 294.30 (83.602) | 312.43 (93.924)
  Week 25: number analyzed (Participants) | 17 | 10 | 93 | 61
  Week 25 | 304.98 (102.934) | 340.71 (72.911) | 315.32 (97.020) | 322.71 (103.865)
Statistical Analysis 1: Comparison: BYM338 70 mg vs Placebo; Test type: Superiority; p = 0.576, Mixed Models Analysis; Mean Difference (Final Values) = -3.32, 95% CI 2-sided [-37.6 to 30.95]
Statistical Analysis 2: Comparison: BYM338 210 mg vs Placebo; Test type: Superiority; p = 0.178, Mixed Models Analysis; Mean Difference (Final Values) = 19.60, 95% CI 2-sided [-22.2 to 61.41]
Statistical Analysis 3: Comparison: BYM338 700 mg vs Placebo; Test type: Superiority; p = 0.163, Mixed Models Analysis; Mean Difference (Final Values) = 10.31, 95% CI 2-sided [-10.4 to 30.98]

3. Secondary Outcome: Change From Baseline to Week 25 in Usual Gait Speed (GS) Over 4 Meters
Description: Change from Baseline to Week 25 in usual Gait speed (GS) over 4 meters Gait speed in this study was assessed as part of the SPPB, over a 4 meter distance of a 6 meter course. This test assessed a person's usual walking speed, which was defined as the speed a person normally walks from one place to another without urgency (e.g., walking down a hallway).
Time Frame: baseline, week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: m/sec
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo
Number analyzed (Participants) | 19 | 18 | 113 | 67
m/sec
  Baseline | 2.37 (0.684) | 2.72 (0.752) | 2.58 (0.624) | 2.70 (0.493)
  Week 25: number analyzed (Participants) | 17 | 10 | 94 | 62
  Week 25 | 3.12 (0.857) | 3.60 (0.699) | 3.30 (0.902) | 3.23 (0.838)
Statistical Analysis 1: Comparison: BYM338 70 mg vs Placebo; Test type: Superiority; p = 0.488, Mixed Models Analysis; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.10 to 0.10]
Statistical Analysis 2: Comparison: BYM338 210 mg vs Placebo; Test type: Superiority; p = 0.055, Mixed Models Analysis; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.02 to 0.22]
Statistical Analysis 3: Comparison: BYM338 700 mg vs Placebo; Test type: Superiority; p = 0.161, Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.03 to 0.09]

4. Secondary Outcome: Percentage Change From Baseline to Week 25 on Appendicular Skeletal Muscle Index (ASMI) Measured by Dual Energy X-ray Absorptiometry (DXA)
Description: Change from Baseline to Week 25 on appendicular skeletal muscle index (ASMI) measured by Dual Energy X-ray Absorptiometry (DXA) Appendicular skeletal muscle index (ASMI) is a core requirement for determining the presence of sarcopenia and is calculated as the sum of the appendicular lean mass (kg) of the two upper and two lower limbs quantified by DXA, divided by height (m^2). Therefore, an increase in ASMI indicates an increase in the quantity of an individual's lean mass.
Time Frame: baseline, week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo
Number analyzed (Participants) | 19 | 18 | 113 | 67
Percent Change
  Baseline | 5.99 (0.886) | 5.87 (0.795) | 5.70 (0.823) | 5.55 (0.753)
  Week 25: number analyzed (Participants) | 16 | 11 | 92 | 62
  Week 25 | 6.04 (0.947) | 6.42 (0.849) | 6.10 (0.836) | 5.60 (0.717)
Statistical Analysis 1: Comparison: BYM338 70 mg vs Placebo; Test type: Superiority; p = 0.213, Mixed Models Analysis; Mean Difference (Net) = 1.01, 95% CI 2-sided [0.99 to 1.03]
Statistical Analysis 2: Comparison: BYM338 210 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.06, 95% CI 2-sided [1.03 to 1.09]
Statistical Analysis 3: Comparison: BYM338 700 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.06, 95% CI 2-sided [1.05 to 1.08]

5. Secondary Outcome: Percentage Change From Baseline to Week 25 on Total Lean Body Mass Measured by Dual Energy X-ray Absorptiometry (DXA)
Description: Change from Baseline to Week 25 on Total lean body mass and appendicular skeletal muscle index (ASMI) measured by Dual Energy X-ray Absorptiometry (DXA) total lean body mass (LBM) is measured by dual energy x-ray absorptiometry (DXA).Percent Change = [(LBM at Visit - LBM at Baseline) / LBM at Baseline] * 100.
Time Frame: baseline, week 25
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo
Number analyzed (Participants) | 19 | 18 | 113 | 67
Percent Change
  Baseline | 37.44 (8.507) | 35.84 (7.300) | 35.39 (8.891) | 33.65 (6.890)
  Week 25: number analyzed (Participants) | 16 | 11 | 92 | 62
  Week 25 | 38.26 (8.660) | 39.52 (8.343) | 37.86 (9.064) | 33.95 (6.921)
Statistical Analysis 1: Comparison: BYM338 70 mg vs Placebo; Test type: Superiority; p = 0.458, Mixed Models Analysis; Mean Difference (Net) = 1.00, 95% CI 2-sided [0.98 to 1.02]
Statistical Analysis 2: Comparison: BYM338 210 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.05, 95% CI 2-sided [1.03 to 1.08]
Statistical Analysis 3: Comparison: BYM338 700 mg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.06, 95% CI 2-sided [1.04 to 1.07]

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for the maximum actual duration of treatment exposure and follow up for a participant per the protocol for approximately 25 weeks.
Arm/Group | BYM338 70 mg | BYM338 210 mg | BYM338 700 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 2/113 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/19 | 3/18 | 14/113 | 5/67
Other Adverse Events (participants affected / at risk) | 12/19 | 13/18 | 94/113 | 41/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 70 mg (N=19) | BYM338 210 mg (N=18) | BYM338 700 mg (N=113) | Placebo (N=67)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Aortic injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 70 mg (N=19) | BYM338 210 mg (N=18) | BYM338 700 mg (N=113) | Placebo (N=67)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1 | 2
Androgen deficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Trichiasis (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 6 | 1
Dental necrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 22 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 8 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 5 | 0
Infusion site swelling (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 1
Oedema (General disorders) | 1 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 6 | 2
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 5 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 5 | 5
Urinary tract infection (Infections and infestations) | 1 | 0 | 6 | 1
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 5 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 5 | 7
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 28 | 24
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 3 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 6 | 0
Liver function test increased (Investigations) | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 5 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 37 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | 3
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 6 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 4 | 0
Headache (Nervous system disorders) | 0 | 0 | 5 | 3
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0 | 3 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-07-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT02333331/SAP_000.pdf
  • Study Protocol (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT02333331/Prot_001.pdf